CLINICAL TRIAL: NCT06077708
Title: Effect of Vitamin D Supplementation in Addition to Non-surgical Periodontal Treatment in Individuals With Type II Diabetes Mellitus and Periodontitis
Brief Title: Diabetes Mellitus and Periodontitis and Vitamin D Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Assoc. Prof., Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/040
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus Type 2 With Periodontal Disease
Keywords: Periodontitis; Type 2 periodontitis; 25(OH)D3; HbA1c
MeSH Terms: conditions — Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D3K2 with periodontal therapy (Active Comparator): Individuals given D3K2 with periodontal therapy were included in the test group.All serum and gingival crevicular fluid samples from individuals who underwent non-surgical periodontal treatment were taken again at 3rd and 6th months, and clinical periodontal measurements were recorded. Glycated hemoglobin A1c (HbA1c), fasting blood glucose (FBG), 25(OH)D3, parathyroid hormone (PTH), calcium (Ca) and magnesium (Mg) values were determined in serum samples. GCF and serum IL-1ß and IL-10 values were analyzed by enzyme-linked immunosorbent analysis (ELISA).
  Interventions: Dietary Supplement: Vitamin D3K2
- Placebo with periodontal therapy (Placebo Comparator): Individuals given placebo with periodontal therapy were included in the control group.All serum and gingival crevicular fluid samples from individuals who underwent non-surgical periodontal treatment were taken again at 3rd and 6th months, and clinical periodontal measurements were recorded. Glycated hemoglobin A1c (HbA1c), fasting blood glucose (FBG), 25(OH)D3, parathyroid hormone (PTH), calcium (Ca) and magnesium (Mg) values were determined in serum samples. GCF and serum IL-1ß and IL-10 values were analyzed by enzyme-linked immunosorbent analysis (ELISA).
  Interventions: Other: Saline Solution

INTERVENTIONS:
Dietary Supplement: Vitamin D3K2 — Non-surgical periodontal treatment was applied to all individuals included in the study. 2 drops of the preparation containing 25 µg D3 [1000 IU] and 11.25 µg K2 in each drop were given per day to participants in the test group.
  Arms: D3K2 with periodontal therapy
Other: Saline Solution — Non-surgical periodontal treatment was applied to all individuals included in the study and saline solution (0.9% NaCl) was given as placebo, 2 drops per day to particiapants in the control group.
  Arms: Placebo with periodontal therapy

SUMMARY:
This study investigates the clinical and biochemical results of vitamin D supplementation in addition to non-surgical periodontal treatment in individuals with Type II diabetes mellitus and periodontitis.

DETAILED DESCRIPTION:
38 individuals with T2DM and periodontitis were included into the study. Clinical periodontal measurements including probing depth, clinical attachment level, plaque and gingival indices were recorded The individuals included in the study were divided into two groups: Individuals given D3K2 with periodontal therapy were included in the test group, and individuals given placebo with periodontal therapy were included in the control group. All serum and gingival crevicular fluid samples from individuals who underwent non-surgical periodontal treatment were taken again at 3rd and 6th months, and clinical periodontal measurements were recorded. Glycated hemoglobin A1c (HbA1c), fasting blood glucose (FBG), 25(OH)D3, parathyroid hormone (PTH), calcium (Ca) and magnesium (Mg) values were determined in serum samples. GCF and serum IL-1ß and IL-10 values were analyzed by enzyme-linked immunosorbent analysis (ELISA).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with Stage I-II periodontitis
2. Individuals with HbA1c value ≥6.5 and diagnosed with type 2 DM according to ADA at least 1 year before the study
3. Individuals who do not have a systemic disease other than DM
4. Individuals who do not have systemic complications of diabetes
5. Individuals with 25(OH)D3 value between 20 ng/mL and 30 ng/mL
6. Individuals who are under the control of a doctor for their diabetes
7. Individuals who have not used any antibiotics or long-term anti-inflammatory drugs in the last 6 months
8. Individuals who have not received periodontal treatment in the last 6 months
9. Individuals with BMI value of 18.5 to 30 kg/m2

Exclusion Criteria:

1. Smokers
2. Individuals who use alcohol
3. Pregnant or lactating individuals
4. Individuals taking any antioxidant or vitamin supplements

Ages: 39 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Biochemical Data | At the first 3 and 6th months post treatment for the test and control groups.
  HbA1c
Periodontal Clinical Parameters | At the 3rd and 6th months post treatment for the test and control groups.
  Probing depth, clinical attachment level

SECONDARY OUTCOMES:
Biochemical Data | At the 3rd and 6th months post treatment for the test and control groups.
  Serum 25(OH)D3 value

CONTACTS AND LOCATIONS:
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No